CLINICAL TRIAL: NCT05329987
Title: Analysis of Postural Transitions in Subjects Affected by Parkinson Disease
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: FDG_PosTrans
Record Dates: First submitted 2022-04-04; First posted 2022-04-15 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Rehabilitation; Postural Transfers
MeSH Terms: conditions — Parkinson Disease | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson Disease: Rehabilitation according to Physiotherapy and Occupational Therapy European Guidelines for Parkinson Disease.
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — Intervention focused on balance, gait and postural transfers rehabilitation. 20 session of 90 minutes (60 minutes of physiotherapy and 30 minutes of occupational therapy), 2 times a week, for 10 weeks.

SUMMARY:
This observational trial aims to evaluate the effect of Rehabilitation on Postural Transfers (PTs) in subjects affected by Parkinson Disease. The PTs are evaluated by an inertial sensor (a device composed by an accelerometer, a gyroscope and a magnetometer) attached to the subjects. The data obtained by the inertial sensor are kinematic (e.g. acceleration and angular speed) and spatiotemporal parameters (e.g. time to completion and velocity). Additional clinical evaluations are carried out at the beginning and end of the rehabilitative intervention.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Idiopathic Parkinson's Disease;
* Subjects should be in a positive therapeutic window or in the ON phase during the evaluations;
* Subjects must be able to walk at least 10 meters independently with or without any walking aid

Exclusion Criteria:

* Non-clinically stable subjects;
* Subjects in OFF phase during the evaluations;
* Other neurological conditions (e.g. stroke, peripheral neuropathies, etc.);
* Other pathologies that can negatively influence the subject's walking ability (e.g. surgery at the lower limbs in the previous 6 months, important deformities at the lower limbs, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of subjects affected by Parkinson Disease
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change in execution time of Postural Transfers | Change from Baseline at 10 weeks
  The execution time is measured via an inertial measurement unit attached to the back of the patient
Change of execution velocity of Postural Transfers | Change from Baseline at 10 weeks
  The execution velocity is measured via an inertial measurement unit attached to the back of the patient. Specifically the velocity are measured as the Root Mean Square of gyroscope signal.
Change of antero-posterior acceleration during Postural Transfers execution | Change from Baseline at 10 weeks
  The antero-posterior acceleration is measured via an inertial measurement unit attached to the back of the patient.
Change of superior-inferior acceleration during Postural Transfers execution | Change from Baseline at 10 weeks
  The superior inferior acceleration is measured via an inertial measurement unit attached to the back of the patient.

SECONDARY OUTCOMES:
Change in Time Up and Go Test | Change from baseline at 10 weeks
Change in 10 meter walking test | Change from baseline at 10 weeks
Change in Berg Balance Scale Score | Change from baseline at 10 weeks
Change in Short-Form 12 score | Change from baseline at 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Buraschi, PT, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi
Locations (1):
- Fondazione Don Carlo Gnocchi, Rovato, BS, Italy

IPD SHARING:
Plan to Share IPD: Undecided